CLINICAL TRIAL: NCT05527496
Title: Effect of Hp Infection on the Quality of Gastric Mucosa Preparation and Study on Different Gastric Mucosa Preparation Schemes in Patients With Hp Infection
Brief Title: Effect of Hp Infection on the Quality of Gastric Mucosa Preparation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: individualliu
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Helicobacter pylori infection: Patients with H. pylori infection identified by testing for H. pylori.
- Patients not infected with Helicobacter pylori: Patients without H. pylori infection identified by H. pylori testing.

SUMMARY:
The purpose of this study was to evaluate the effect of Helicobacter pylori infection on the quality of gastric mucosa preparation.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effect of Helicobacter pylori infection on the quality of gastric mucosa preparation by comparing the cleanliness of gastric mucosa between patients with Helicobacter pylori infection and those without Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults who volunteered to participate in this study and signed an informed consent form
* Have been tested for Helicobacter pylori and have definite test results

Exclusion Criteria:

* Contraindications for gastroscopy (such as severe cardiopulmonary diseases, liver and kidney dysfunction, shock, etc.)
* History of upper gastrointestinal surgery
* Therapeutic endoscopy and emergency surgery are required
* Recent history of upper gastrointestinal bleeding
* Corrosive substance ingestion
* The pregnancy
* Abnormal mental state cannot cooperate with the examination
* Patients with contraindications to the drugs used in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All outpatients or inpatients requiring general gastroscopy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Cleanliness of gastric mucosa | The time the patient underwent gastroscopy procedure
  The visibility of gastric mucosa was scored for four parts of the stomach (antrum, upper body, lower body and fundus).

SECONDARY OUTCOMES:
Time to complete gastroscopy | The day of gastroscopy
  The time from the start of the endoscopy to the complete removal of the endoscope
Patient comfort score | Records were made on the 1 day of the gastroscopy
  Prior to endoscopy, the patient was instructed to indicate the level of discomfort on a visual analogue scale, which was rated by the patient on a scale of 0 to 10, with 0 indicating no discomfort and 10 indicating maximum discomfort.
adverse reaction | Within 24 hours after endoscopy
  Adverse reactions to study drugs, and respiratory, cardiovascular, or endoscopic adverse events.
Endoscopic findings | About 15 days after endoscopy
  The diagnostic results were recorded under gastroscopy, and if the biopsy was taken under gastroscopy, the pathological results were also recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No